CLINICAL TRIAL: NCT06834386
Title: A Pilot Randomized, Open Label Trial of Orexin Receptor Antagonist for Insomnia in Hospitalized Patients With Cancer to Prevent Delirium
Brief Title: Suvorexant for Insomnia to Prevent Delirium in Hospitalized Cancer Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-005893; NCI-2025-00771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-005893 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Solid Neoplasm; Delirium; Hematopoietic and Lymphatic System Neoplasm; Insomnia
MeSH Terms: conditions — Delirium; Sleep Initiation and Maintenance Disorders | interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic; suvorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (suvorexant, standard of care) (Experimental): Patients receive suvorexant PO QD at bedtime and standard of care for hospital associated insomnia for 3-7 days in the absence of unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Interview; Other: Questionnaire Administration; Drug: Suvorexant
- Arm II (standard of care) (Active Comparator): Patients receive standard of care for hospital associated insomnia for 3-7 days in the absence of unacceptable toxicity.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Drug: Suvorexant — Given PO
  Other Names: Belsomra; MK-4305
  Arms: Arm I (suvorexant, standard of care)

SUMMARY:
This phase IV trial compares suvorexant with standard of care to standard of care alone for improving difficulty sleeping (insomnia) and reducing confusion (delirium) in hospitalized cancer patients. Delirium can lengthen hospitalization, increase the delay of cancer treatment and can even increase the risk of premature death. Suvorexant is in a class of medications called orexin receptor antagonists. It works by blocking the action of a certain natural substance in the brain that causes wakefulness. Giving suvorexant with standard of care to treat insomnia may be more effective compared to standard of care alone in reducing the development of delirium in hospitalized cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Feasibility of a subsequent full scale randomized clinical trial (RCT) conducted at Mayo Clinic using the same methodology as outlined in this protocol (as this study is a pilot).

SECONDARY OBJECTIVE:

I. To generate preliminary data to determine if inpatient standard of care (i.e. sleep enhancement) is followed in both a study arm receiving standard of care alone and one receiving standard of care plus suvorexant.

EXPLORATORY OBJECTIVES:

I. To collect preliminary data to investigate the hypotheses that use of suvorexant in addition to standard of care for hospitalized adults with cancer will result in a decreased incidence of delirium, increased time to onset of delirium, and decreased number of delirium days in hospital as compared to standard of care alone.

II. To build a data collection and analysis infrastructure for a full scale RCT at Mayo Clinic if feasibility is demonstrated.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive suvorexant orally (PO) once daily (QD) at bedtime and standard of care for hospital associated insomnia for 3-7 days in the absence of unacceptable toxicity.

ARM II: Patients receive standard of care for hospital associated insomnia for 3-7 days in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Presence of advanced active malignancy and insomnia despite nonpharmacologic management
* Anticipated hospital course of at least 3 days post randomization as judged by the patient's primary inpatient team
* One or more of the following risk factors of delirium:

  * Age 75 or above
  * Hearing impairment
  * Vision impairment
  * Initiation of 8 or new medications since start of hospitalization
  * Chronic kidney disease III or greater
  * Congestive heart failure
  * Hospitalization for 14 or more days
  * Dehydration requiring ongoing use of intravenous (IV) hydration
  * Electrolyte imbalance requiring ongoing correction

Exclusion Criteria:

* Inability to consent
* Current pregnancy
* Women of childbearing potential (defined as women under age 55 without a personal history of surgical or chemotherapy-induced sterility)
* Current or prior delirium in the active hospitalization
* Concurrent use of strong/moderate CYP3A4 inducers and inhibitors (including but not limited to -azole antifungals, amiodarone, phenytoin, carbamazepine, etc.)
* Use of any benzodiazepine, benzodiazepine receptor modulator, or first generation antihistamine class medication within 72 hours prior to enrollment
* Personal history of narcolepsy
* Personal history of other primary sleep disorders including obstructive sleep apnea
* Personal history of alcohol use disorder
* Personal history of substance use disorder
* Personal history of cirrhosis
* Transaminitis more than 3 times the upper limit of normal
* History of obstructive lung disease other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Recruitment | Up to 1 year
  Feasibility will be defined as the ability to recruit 14 patients to the study with 20% or less study attrition.

SECONDARY OUTCOMES:
Adherence to standard of care | Baseline (enrollment), assessed 3-7 days while in the hospital or until discharged, whichever comes first
  Adherence to standard of care will be compared within each arm and between arms. Will be monitored with adequate adherence being defined as at 5/7 patients in each group and a between-group difference of no more than 2.
Change in Insomnia Severity Index score | Baseline (enrollment), assessed 3-7 days while in the hospital or until discharged, whichever comes first
  Reduction of at least two points will be defined as clinical improvement. The Insomnia Severity Index consists of 7 items related to current (i.e., last 2 weeks0 severity of insomnia problems. Three items are rated on a scale of 0-4 where 0=none; 1=mild; 2=moderate; 3=severe; and 4=very severe. The remaining items are answered on similar scales of 0-4 (e.g., 0=not at all; 1=a little; 2=somewhat; 3=much; 4=very much).

CONTACTS AND LOCATIONS:
Overall Officials: Regina M. Mackey, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials